CLINICAL TRIAL: NCT07360639
Title: Effectiveness of a Combination Cream of Gayo Arabica Coffee Bean Extract and Aceh Patchouli (Pogostemon Cablin Benth) Compared to Urea Cream for Dry Skin
Brief Title: The Effectiveness of Herbal Creams Compared to Urea in Dry Skin Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitas Syiah Kuala (Other)
Responsible Party: Principal Investigator, Wahyu Lestari, Associate Professor, Universitas Syiah Kuala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192/ETIK-RSUDZA/2025
Record Dates: First submitted 2026-01-11; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Dry Skin; Xerosis Cutis
Keywords: Coffee; patchouli; xerosis; antioxidant; herbal
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- safety check subject (Active Comparator): this subject receive cream combination of Gayo Arabica coffee husk extract and Aceh patchouli as patch test to test the safety of this cream combination. The result was documented at 48 hours, 72 hours, and 96 hours after patch application and assessed using International Contact Dermatitis Research Group standard
  Interventions: Drug: combination cream
- experimental group (Active Comparator): this group received cream combination of Gayo Arabica coffee husk extract and Aceh patchouli to be applied at the dry skin. The cream applied twice daily. Assessment was done at 6 weeks after cream application
  Interventions: Drug: combination cream
- Control group (Other): this group received cream containing 10% urea to be applied at the dry skin. The cream applied twice daily. Assessment was done at 6 weeks after cream application
  Interventions: Drug: control cream

INTERVENTIONS:
Drug: combination cream — cream containing gayo arabica coffee husk extract and aceh patchouli extract was made. The cream formulation method was taken from previous research
  Arms: experimental group; safety check subject
Drug: control cream — this intervention was application of cream containing 10% urea as the standard method in treatment of xerosis cutis
  Arms: Control group

SUMMARY:
The goal of this Clinical trial is to Determine the effectiveness of a cream combining Gayo Arabica coffee bean extract and Aceh patchouli compared to urea cream for dry skin in Patients with dry skin, aged 18-65 years old who meet the inclusion criteria. The main question it aims to answer is:

Can cream combination of Gayo Arabica coffee husk extract and Aceh patchouli be used on humans? is cream combination of Gayo Arabica coffee husk extract and Aceh patchouli clinically effective in improving dry skin

Researchers will compare cream combination of Gayo Arabica coffee bean extract and Aceh patchouli to 10% urea cream see the better outcome.

Participants will apply the cream corresponding to their group for twice a day for 6 weeks.

DETAILED DESCRIPTION:
Coffee husks and patchouli are local plants in Aceh that contain high levels of antioxidants and are believed to help moisturize and repair the skin. Previous research, both in silico and in vivo, found that the combination of Arabica coffee bean skin and patchouli extracts is safe to use and has the ability to inhibit the skin aging process. Therefore, testing and verification are needed for clinical trials of this cream on humans with dry skin. Based on the background of the problem described above, the problem can be formulated as is cream combination of Gayo Arabica coffee husk extract and Aceh patchouli clinically safe and effective in improving dry skin, increasing skin hydration, reducing ODSS scores and water loss levels, and improving patients' quality of life (DLQI) compared to 10% urea cream in patients at RSUDZA? The safety of cream combination of Gayo Arabica coffee husk extract and Aceh patchouli was tested on healthy individuals using patch tests. Research subjects were selected using purposive sampling, according to the inclusion criteria. The phase 2 study design was a randomized controlled trial (RCT) using a double-blind method to compare cream combination of Gayo Arabica coffee husk extract and Aceh patchouli with 10% urea cream. The study was conducted at Dr. Zainoel Abidin Hospital (RSUDZA), with subjects being patients with dry skin, aged 18-65 years, using consecutive sampling, with a total of 64 subjects (32 per group) + 10% of the total subjects (total 70 subjects) and according to the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years old
* Diagnosed with xerosis cutis
* not using any moisturizer for more than 2 weeks
* dry skin at extremity

Exclusion Criteria:

* no history of coffee, patchouli, urea, or cream composition allergy
* secondary infection lession appeared
* pregnant or breastfeeding woman
* history of using another topical drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
herbal cream effectiveness in treating dry skin | 6 weeks
  this outcome was assessed the effectiveness of the cream by using overall dry skin score (ODSS) and the difference value of transepidermal water loss (TEWL). this assessment was carried out using physiological change such as scaling, itching, pain, erythema, and fissures. The water loss was assessed in the unit of grams per square meter per hour (g/m²/h)
the safety assessment of herbal cream application on human skin | 96 hours after cream application
  the cream safety was assessed using international contact dermatitis research group (ICDRG) standard. this tool graded the physiological change based on the lesion that appeared.

CONTACTS AND LOCATIONS:
Locations (1):
- dr. Zainoel Abidin General Hospital, Banda Aceh, Nanggore Aceh Darussalam, Indonesia

IPD SHARING:
Plan to Share IPD: No
IPD will not (or might not) be shared due to ethical considerations, data ownership restrictions, and the need to protect participant confidentiality, as the data are sensitive and collected under informed consent that limits secondary use

REFERENCES:
- [Background] Lestari W, Hasballah K, Listiawan MY, Sofia S. Metabolite Signature of Fresh and Long-term Stored Coffee Pulp and Husk. Makara J Sci [Internet]. 30 September 2022;26(3).
- [Background] Paradila ED, Prasetya F, Almeida M. Formulasi Sediaan Krim Body scrub dari Serbuk Kopi yang Dikombinasikan dengan Minyak Zaitun sebagai Pencerah dan Pelembab Kulit. Proceeding Mulawarman Pharm Conf [Internet]. 31 Mei 2022;15:48-52.
- [Background] Lestari W, Dewi Ismida F, Hajar S, Clarissa Namiko R. The Effect of Combination Cream of Patchouli Extract and Arabica Gayo Coffee Peel Extract on Aging Skin. Berk Ilmu Kesehat Kulit dan Kelamin [Internet]. 31 Juli 2024;36(2):113-22.